CLINICAL TRIAL: NCT04792073
Title: A Phase II Single-Arm Clinical Trial Assessing Comprehensive Ablative Radiation Therapy With Avelumab in Unresectable and Metastatic Merkel Cell Carcinoma (CARTA)
Brief Title: Study of Avelumab and/or Radiation Therapy in People With Advanced Merkel Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-195
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Merkel Cell Carcinoma
Keywords: unresectable; metastatic; stage III; stage IV; Comprehensive Ablative Radiation Therapy; Avelumab; 20-195
MeSH Terms: conditions — Carcinoma, Merkel Cell; Neoplasm Metastasis | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: A Phase II Single-Arm Clinical Trial Assessing Comprehensive Ablative Radiation Therapy with Avelumab in Unresectable and Metastatic Merkel Cell Carcinoma (CARTA)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avelumab and Radiation Therapy (Experimental): Will receive avelumab at the FDA approved dose and schedule of 800 mg IV over 60 minutes (+20 minutes / -10 minutes) every 2 weeks (+/- 3 days) until treatment intolerance or disease progression occurs or 2 years of study therapy have been administered; standard of care Avelumab therapy after 2 years is permitted. Comprehensive Ablative Radiation Therapy (CART) will be initiated between the first and second dose of Avelumab. Comprehensive ablative radiation therapy will be given according to guidelines.
  Interventions: Drug: Avelumab; Radiation: Comprehensive Ablative Radiation Therapy

INTERVENTIONS:
Drug: Avelumab — Avelumab 800 mg given intravenously over 60 minutes (+20 minutes / -10 minutes) every 2 weeks (+/- 3 days)
Radiation: Comprehensive Ablative Radiation Therapy — Comprehensive ablative radiation therapy 24 Gy in 3 fractions every 2-3 days

SUMMARY:
This study will test the use of comprehensive ablative radiation therapy (CART), with the immunotherapy drug avelumab, in people with Merkel cell carcinoma (MCC) that has progressed after treatment and cannot be removed with surgery. The study researchers want to find out if CART works well when combined with avelumab.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Merkel cell carcinoma which is unresectable or metastatic, stage III or IV
* Prior first-line treatment with aPD1 monotherapy (defined as at least one dose of pembrolizumab, avelumab, nivolumab, etc.) with evidence of progression of disease ≥10 weeks after starting therapy, in the absence of significant clinical deterioration

  * Patients with clinical deterioration during aPD1 monotherapy are eligible ≥6 weeks after starting aPD1 therapy
  * Criteria for clinical deterioration to be determined and agreed upon by treating physician and Principal Investigator
* All detectable sites of MCC are amenable to comprehensive ablative radiation therapy in opinion of treating radiation oncologist and principal investigator
* ≥18 years of age
* Performance status ≤2 on the Eastern Cooperative Oncology Group Performance Scale
* Able to provide valid written informed consent
* Normal organ and marrow function

  * Hematologic: Neutrophil count ≥1500/mm^3, platelet count ≥100,000/mm^3, hemoglobin ≥9 g/dL
  * Hepatic: Total bilirubin ≤ 1.5 times the upper limit of normal, unless Gilbert's syndrome; aspartate transaminase and alanine transaminase ≤ 2.5 times the upper limit of normal (in the absence of hepatobiliary metastases); ≤ 3.0 times the upper limit of normal (in the presence of hepatobiliary metastases)
  * Renal: Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula.

Exclusion Criteria:

* Prior systemic therapy for MCC other than first-line aPD1 monotherapy (ie, chemotherapy)
* Pregnancy or breastfeeding
* Adverse events due to prior cancer therapy which are grade 3 or higher and have not resolved

  °Patients with prior grade 3 or higher immune related adverse events are not eligible, even if they have resolved
* Prior severe hypersensitivity reaction (CTCAE version 5.0 grade ≥3) to avelumab
* Prior radiotherapy which precludes the ability to safely deliver comprehensive ablative radiation therapy in the opinion of the treating radiation oncologist and principal investigator

  °Institutional guidelines for reirradiation will be used when making this determination
* Known central nervous system metastases
* Known clinically significant cardiovascular disease, defined as:

  * Stroke or myocardial infarction within 6 months of first dose of avelumab
  * Symptomatic congestive heart failure (New York Heart Association Class 2 or higher)
  * Serious arrhythmia requiring anti-arrhythmic agents
* Known Human Immunodeficiency Virus infection
* Known Hepatitis B or C infection requiring ongoing treatment
* Vaccination within 4 weeks of first dose of avelumab

  °Inactivated vaccines are permissible
* Iatrogenic immunosuppression with daily systemic corticosteroid equivalent of >10 mg of prednisone
* Active autoimmune disease that may cause clinical deterioration during immunotherapy

  °Including, but not limited to:
* Inflammatory bowel disease or immune colitis
* Immune mediated pneumonitis or pulmonary fibrosis
* History of solid organ or hematopoietic transplant
* Active infection requiring systemic therapy
* Active suicidal ideation or behavior
* Comorbid or diagnostic abnormalities which would interfere with interpretation of study results
* Known hematopoietic cancer or dysfunction (i.e., leukemia, lymphoma)
* Known non-MCC solid tumor with known metastasis or estimated risk of metastasis >20% within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
progression free survival | at 12 weeks
  measured by RECIST 1.1

SECONDARY OUTCOMES:
overall response rate | up to 12 weeks
  measured by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Christoper Barker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm